CLINICAL TRIAL: NCT04147221
Title: An Open-label Pharmacokinetic Study of Imipenem-Relebactam in Critically Ill Patients With Augmented Renal Clearance
Brief Title: Imipenem-Relebactam Pharmacokinetics in Augmented Renal Clearance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HHC-2019-0237
Record Dates: First submitted 2019-10-29; First posted 2019-11-01 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Sepsis
Keywords: beta-lactam; pharmacokinetics
MeSH Terms: conditions — Sepsis | interventions — imipenem, cilastatin and relebactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imipenem-Relebactam (Experimental): Participants will receive a single dose of intravenous imipenem-relebactam (500mg-250mg) as a 30 minute infusion.
  Interventions: Drug: Imipenem-relebactam

INTERVENTIONS:
Drug: Imipenem-relebactam — After receipt of imipenem-relebactam, participants will have six blood samples collected over 6 hours for determination of imipenem and relebactam concentrations.

SUMMARY:
Critically ill patients with sepsis undergo several physiological alterations that can alter the distribution, metabolism, and elimination of drugs. Some patients with sepsis may realize enhanced cardiac output leading to increases in glomerular filtration that result in increasing drug clearance. This clinical state is referred as Augmented Renal Clearance (ARC). Importantly, many beta-lactam antibiotics can be adversely affected by ARC, and some of these agents required increasing dosage to compensate for enhanced clearance. Imipenem-relebactam is a new broad spectrum antibiotic. This study is designed to assess the pharmacokinetics of both components, imipenem and relebactam, in critically ill patients with ARC.

DETAILED DESCRIPTION:
This is a single center, open-label study to determine imipenem-relebactam pharmacokinetics in critically ill patients with Augmented Renal Clearance (ARC). Twelve patients with suspected ARC will be enrolled to ensure complete pharmacokinetic data in at least eight patients with confirmed ARC. Confirmation of ARC will be established by eight hour urine creatine determination. Each participant will receive a single dose of imipenem-relebactam (500mg/250mg) followed by six blood samples over a 6 hour interval to determine concentrations. Non-compartmental and population pharmacokinetic analyses will be determined to assess the effects of ARC on imipenem and relebactam pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* APACHE II score > 12 and ≤ 35;
* Creatinine clearance (CrCL) ≥150 mL/min (as calculated by the Cockcroft-Gault equation using ideal or adjusted body weight) within 24 hours of dosing;
* Documented infection or presumed infection as confirmed by the presence of at least one of the following criteria within the past 72 hours:

  1. Documented fever (oral, rectal, tympanic, or core temperature > 38.5° C)
  2. Hypothermia (oral, rectal, tympanic, or core temperature < 35.0° C)
  3. An elevated white blood cell (WBC) count ≥ 12,000 cells/mm3

Exclusion Criteria:

* If female, currently pregnant or breast feeding;
* History of any moderate or severe hypersensitivity or allergic reaction to any β-lactam antibiotic (Note: mild rash or erythema to penicillin or cephalosporin antibiotics would not disqualify a patient if they have received a carbapenem without problem);
* History of chronic kidney disease, hemodialysis, or peritoneal dialysis; or history of acute renal replacement therapy (e.g., hemodialysis, hemofiltration, hemodiafiltration) or extracorporeal membrane oxygenation (ECMO) associated with current illness;
* Suspected rhabdomyolysis or creatine kinase > 10,000 U/L;
* Any serum creatinine (SCr) before dosing that is increased ≥ 0.3 mg/dL from the baseline SCr used qualifying for enrollment;
* Urinary output <20 ml/hour for at least 2 hours (oliguria) within 24 hours before enrollment;
* Sustained (at least 1 hour) hypotension (systolic pressure < 90 mmHG or mean arterial pressure < 55 mmHg) refractory to vasopressors or intravenous fluid resuscitation for at least 24 hours before enrollment;
* Significant anemia defined as a hemoglobin < 8 g/dL at baseline;
* Use of probenecid, valproic acid, or imipenem within 3 days before study drug infusion;
* Acute liver injury, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times the upper limit of normal, or AST or ALT > 3 times the upper limit of normal with an associated total bilirubin > 2 times upper limit of normal;
* Any rapidly-progressing disease or immediately life-threatening illness (defined as imminent death within 48 hours in the opinion of the investigator);
* Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the patient or the quality of study data;
* Planned or prior participation in any other interventional drug study within 30 days.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Kuti, PharmD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imipenem-Relebactam
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Nine critically-ill patients or their next-of-kin consented to participate in this single-center, open-label, pharmacokinetic study. One patient was excluded from the pharmacokinetic analyses after enrollment due to loss of vascular access thereby preventing blood sample collection.
Arm/Group | Imipenem-Relebactam
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 8
Total Body Weight [Mean (Standard Deviation); unit: kg] | 89 (16)
APACHE II Score [Mean (Standard Deviation); unit: scores on a scale] — The APACHE II (Acute Physiology and Chronic Health Evaluation II) Score evaluates the severity of illness in critically ill patients based on several physiological parameters, chronic health conditions, and age. The scale ranges from 0-71. The higher the score, the more severe illness and higher risk of mortality.
  scores on a scale | 16 (6)
Cockcroft-Gault CrCL [Mean (Standard Deviation); unit: mL/min] — This metric estimates glomerular filtration (i.e., Creatinine Clearance, ml/min) based on measured serum creatinine, age, weight and sex of the patient (Cockroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. https://pubmed.ncbi.nlm.nih.gov/1244564/).
  mL/min | 193 (62)
Urine Measured CrCL [Mean (Standard Deviation); unit: mL/min] — Description: This metric is measured glomerular filtration (i.e., Creatinine Clearance (CrCL), ml/min) based measured serum and urine creatinine and volume of urine collected over an 8 hour interval. It is calculated as Measured CrCL (ml/min) = (urine creatinine (mg/dL) x urine volume (mL)) / (serum creatinine (mg/dL) x 8 (hours)).
  mL/min | 156 (37)
Albumin [Mean (Standard Deviation); unit: mg/dL] | 2.8 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Imipenem Clearance
Description: The clearance in liters/hour of imipenem from the plasma of critically ill patients with augmented renal clearance
Time Frame: 6 hours [Timepoints taken at 0 hour (within 30 minutes prior to the start of infusion), 0.5 hours (end of infusion), 0.75, 1, 2, 4, and 6 hours after the start of the infusion]
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Imipenem-Relebactam
Number analyzed (Participants) | 8
L/h | 17.31 (5.67)

2. Primary Outcome: Relebactam Clearance
Description: The clearance in liters/hour of relebactam from the plasma of critically ill patients with augmented renal clearance
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Imipenem-Relebactam
Number analyzed (Participants) | 8
L/h | 11.51 (4.79)

3. Secondary Outcome: Imipenem Area Under the Curve (AUC)
Description: The AUC in milligram*hour/liter of imipenem calculated from concentrations collected between zero-6 hours and then extrapolated to infinity
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Imipenem-Relebactam
Number analyzed (Participants) | 8
mg*h/L | 32.33 (11.60)

4. Secondary Outcome: Relebactam Area Under the Curve (AUC)
Description: The AUC in milligram*hour/liter of relebactam calculated from concentrations collected between zero-6 hours and then extrapolated to infinity
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Imipenem-Relebactam
Number analyzed (Participants) | 8
mg*h/L | 25.54 (10.21)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 24 hour window, from the first (and only) imipenem-relebactam dose (0 hour) to the end of blood sampling (6 hours), plus an 18 hour observation window after the last sample was collected, culminating with physical exam. Note: 9 subjects were enrolled and received imipenem-relebactam. Although only 8 subjects were included in results analysis due to inability to obtain blood samples in 1 subject, all 9 subjects are included in the adverse event reporting.
Description: Adverse event - any pathologic or unintended change in the structure (signs), function (symptoms), or chemistry (laboratory values) of the body associated with the use of the study drug, whether or not considered drug related: MILD - present, but easily tolerated MODERATE - discomfort that interferes with usual activities SEVERE - incapacitating, inability to work or do usual activities
Arm/Group | Imipenem-Relebactam
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imipenem-Relebactam (N=9)
Bradycardia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT04147221/Prot_SAP_000.pdf